CLINICAL TRIAL: NCT06542237
Title: Open Label Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Repeated Daily Oral Dosing of YCT-529 for 28 Days or 90 Days in Healthy Men. Healthy Men
Brief Title: Open Label, Repeat Dose Study Evaluating YCT-529 in Healthy Males
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: YourChoice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: YCT-529-02
Record Dates: First submitted 2024-07-03; First posted 2024-08-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Male Contraception
Keywords: male; non-hormonal; male contraception; healthy males; sperm count reduction; sperm motility; impaired spermatogenesis; impaired motility; orally administered; men; vasectomy; awaiting vasectomy; children; father; family planning
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: The study consists of 3 parts: a 28-day Phase 1b part (Part 1), a 90-day Phase 1b part (Part 2) and a 90-day Phase 2a part (Part 3). All participants will receive YCT-529.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YCT-529 (Experimental): Open label, ascending dose, 3 part study (Phase 1b includes Part 1 and 2; and the Phase 2a portion of the study represents Part 3)
  Interventions: Drug: YCT-529

INTERVENTIONS:
Drug: YCT-529 — In the Phase 1b portion of the study (Part 1), 4 dosing cohorts and one optional 5th cohort with 4 participants in each cohort will be evaluated (approximately 20 participants): 15, 30, 90 and 180 mg.
  In the Phase 1b portion of the study (Part 2), 4 dosing cohorts with 4 participants in each cohort will be evaluated (approximately 16 participant): dose to range from 30 mg upto 180 mg.
  In the Phase 2a portion of the study (Part 3), up to 3 cohorts of up to 10 participants (approximately 30 participants) will receive doses within the range of doses that was well tolerated and had biological activity in the Phase 1b portion.

SUMMARY:
This is an open-label, 3 part-study, 28-day or 90-day dose study of YCT-529 in healthy males who have decided to have a vasectomy and are waiting for the procedure and for men who have decided not to father children in the future. The study is aimed at evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics and to assess sexual function and mood.

DETAILED DESCRIPTION:
This is a Phase 1b/2a, multicenter, open label, 28-Day and 90-Day repeat-dose escalation study of YCT-529 in healthy men to evaluate the safety, tolerability, PK and PD, and to assess sexual function and mood. Cohorts will be dosed in the fasted or fed state. In the Phase 1b portion of the study (Part 1), 4 dosing cohorts and one optional 5th cohort with 4 participants each will be evaluated. All participants will receive YCT-529 for 28-days.

In the 1b portion of the study (Part 2), up to 4 dosing cohorts with 4 participants each will be evaluated and will receive YCT-529 for 90-Days. All dose levels will be at or below a dose that was deemed safe and well tolerated upon 28-day administration in Part 1. In the Phase 2a portion (Part 3), up to 3 cohorts will receive doses within the range of doses that was well tolerated and had biological activity in the Phase 1b portion. Each Phase 2a cohort will have up to 10 participants. All participants will receive YCT-529.

The study population in both parts of the study will include healthy men who have decided to have a vasectomy and are waiting for the procedure and men who, in the opinion of the investigator, have made a firm decision not to father children in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in good health as confirmed by physical examination, medical history, and clinical laboratory tests.
2. Participant must provide written informed consent.
3. Participant must be willing and able to communicate and participate in the whole study.
4. Participant is 28 to 70 years of age (inclusive) at the time of consent.
5. Participant has decided to have a vasectomy and is waiting for the procedure or participant, in the opinion of the investigator, has made a firm decision not to father children in the future.
6. Participant has a body mass index (BMI) 18.0 to 35.0 kg/m2.
7. Participant has no history of hormonal therapy or 5-alpha reductase inhibitors use in the 90 days prior to the first screening visit.
8. Participant with partner(s) of childbearing potential agrees to use a method of contraception that is highly effective with any partner (i.e., total abstinence or at a minimum, barrier method plus additional method of contraception) during the study until 28 days after the last dose (Day 56 [Part 1] or Day 118 [Parts 2 and 3]). Condom use is required during the course of the study with partner(s) of both childbearing and non-childbearing potential until Day 56 (Part 1) or Day 118 (Parts 2 and 3) to avoid potential secondary transmission of study drug and ensure the safety of the participants' sexual partner(s). Total abstinence from intercourse during the course of the study until Day 56 (Part 1) or Day 118 (Parts 2 and 3) is considered an acceptable form of contraception if this is in line with participant's preferred and/or usual lifestyle. Condom use is not required while practicing total abstinence.
9. Participant will refrain from donating blood or plasma during the study.
10. Participant will not use cannabis or any other recreational drugs for at least 30 days before the Screening visit and during the study. The marijuana/cannabis test can be positive at Screening but needs to be negative at admission (Day -1) for a volunteer to be eligible for inclusion in the study.
11. Part 1: In the opinion of the investigator, participant is able to adhere to the study requirements, restrictions, schedule of assessments, and requirements related to sperm sample collection and maintenance of the sexual activity diary. Parts 2 and 3: In the opinion of the investigator, participant is able to adhere to the study requirements, restrictions, schedule of assessments, and requirements related to semen sample collection and maintenance of the electronic dosing diary.
12. Part 1: Participant providing at least 2 semen samples during the screening period with sperm parameters within at least the 5th percentile of the WHO range of normality (WHO, 2010 and WHO, 2021):

    * 15 million sperm cells/mL
    * 39 million sperm cells/total ejaculate
    * 40% total motility
    * 30% progressive motility Parts 2 and 3: Participant providing at least 2 semen samples during the screening period with ≥ 15 million sperm cells/mL (at least the 5th percentile of the WHO range of normality [WHO, 2021]).

Exclusion Criteria:

1. Men participating in another clinical study involving an investigational drug within the last 30 days prior to the first dosing or less than 5 elimination half-lives prior to first dosing, whichever is longer.
2. Clinically significant abnormal physical and/or laboratory findings at Screening
3. Abnormal serum chemistry values at screening or admission, that indicate liver or kidney dysfunction or that may be considered clinically significant as determined by the PI, except for bilirubin >20 μmol/L and ALT, AST, GGT and ALP 2-fold above the upper limit of normal. Volunteers with known Gilbert's syndrome will be excluded if total bilirubin is ≥1.5 x ULN.
4. Evidence of renal impairment at screening
5. Use of androgens and selective androgen receptor modulators (SARMs) within 90 days before first screening visit.
6. Volunteers with a body weight < 55 kg.
7. Systolic blood pressure (BP) >140 mmHg (<45 years) or >160 mmHg (≥45 years) and diastolic BP >90 mmHg at screening and admission.
8. Clinically significant abnormal electrocardiogram (ECG) or a duration of corrected QT interval using Bazett's and Fridericia's QT correction methods in ECG (QTc) interval of >450 msec at screening or predose.
9. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease or multiple endocrine deficiencies.
10. Known history of significant cardiovascular, renal, hepatic (cholecystectomy is not permitted), or prostatic disease. Gilbert's syndrome is allowed (volunteer with known Gilbert's syndrome will be excluded if total bilirubin is ≥1.5 x ULN). If volunteer has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (i.e., direct bilirubin <35% of the total bilirubin).
11. Current or clinically relevant history of any psychiatric disorder or clinical assessment of significant suicidal risk or risk of self-injury as per the Investigator's judgement.
12. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients.
13. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Seasonal allergies (e.g., hay fever) are allowed unless considered clinically significant by the investigator.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results at screening visit.
15. Known or suspected alcoholism or drug abuse within the last 2 years that may affect metabolism/transformation of steroid hormones or study treatment compliance.
16. Volunteers who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator or delegate at screening.
17. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type.
18. Current smokers who have consumed at least 5 cigarettes or equivalent amount of nicotine per week within the last 3 months prior to Screening.
19. Confirmed positive drugs of abuse test result at Screening and admission and/or positive marijuana/cannabis test at admission (Day -1).
20. Participants and volunteers who are taking, or have taken, any prescribed or over-the-counter drug or vitamins/herbal remedies/supplements (other than up to 4 g of paracetamol or up to 3.2 g of ibuprofen per day during the 14 days before IMP administration). COVID-19 vaccines are accepted concomitant medications. Other concomitant medications may be accepted at the discretion of both the PI and the Sponsor. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no PD activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardize the safety of the trial participant; and if the use of medication is not considered to interfere with the objectives of the study.
21. Male volunteer with pregnant or lactating partner(s).
22. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.
23. Any other medical condition that, in the opinion of the investigator, could alter the volunteer's well-being, the study conduct, or the interpretability of the results.

    -

Ages: 28 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male participants only
Enrollment: 66 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and nature of any adverse events, dose-limiting adverse events and serious adverse adverse events. | Baseline to 360 days for subjects participating in Parts 1b and 2a
  Assessment of the number and type of adverse events, dose-limiting adverse events and serious adverse events following dosing.
Vital signs assessment (heart rate) | Baseline to Day 360
  Changes from pre-dose values (beats per minute)
Vital signs assessment (blood pressure) | Baseline to Day 360
  Changes from pre-dose values (mm hg)
Vital signs assessment (oral temperature) | Baseline to Day 360
  Changes from pre-dose values (temperature in celsius degrees)
12-lead ECG assessment (heart rate) | Baseline to Day 360
  Changes from pre-dose values (beats per minute)
12-lead ECG assessment (QT interval) | Baseline to Day 360
  Changes from pre-dose values for QT internal length (msec)
12-lead ECG assessment (QTcF Interval) | Baseline to Day 360
  Changes from pre-dose values for QTcF interval length (msec)
12-lead ECG assessment (PR Interval) | Baseline to Day 360
  Changes from pre-dose values for PR interval length (msec)
12-lead ECG assessment (QRS Duration) | Baseline to Day 360
  Changes from pre-dose values for QRS duration (msec)
Clinical laboratory assessment- Hemoglobin Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for hemoglobin (gm/dl)
Clinical laboratory assessment- Hematocrit Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for hematocrit (%)
Clinical laboratory assessment- Packed Cell Volume Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for packed cell volume (%)
Clinical laboratory assessment- Red Blood Cell Sample Test | Baseline to Day 360
  Change from pre-dose value for red blood cells (g/dL)
Clinical laboratory assessment- Mean Corpuscular Volume Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for mean corpuscular volume (fL)
Clinical laboratory assessment- Mean Corpuscular Hemoglobin Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for mean corpuscular hemoglobin (MCH)
Clinical laboratory assessment- Mean Corpuscular Hemoglobin Concentration Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for mean corpuscular hemoglobin concentration (g/dL)
Clinical laboratory assessment- Platelet Count Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for platelets (microL)
Clinical laboratory assessment- White Blood Cell Sample Test | Baseline to Day 360
  Change from pre-dose value for White blood cells (cells/L)
Clinical laboratory assessment- Neutrophil Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for Neutrophils (cells/L)
Clinical laboratory assessment- Lymphocyte Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for Lymphocytes (cells/mcL)
Clinical laboratory assessment- Monocyte Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for Monocytes (cells/L)
Clinical laboratory assessment- Eosinophil Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for Eosinophils (%)
Clinical laboratory assessment- Basophil Blood Sample Test | Baseline to Day 360
  Change from pre-dose value for Basophils (%)
Clinical laboratory assessment- Coagulation Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Prothrombin time (seconds)
Clinical laboratory assessment- Activated Partial Thromboplastin Time Blood Sample Test | Baseline to Day 360
  Changes from pre-dose values for Activated partial thromboplastin time (seconds)
Clinical laboratory assessment- Fibrinogen Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Fibrinogen (mg/dL)
Clinical laboratory assessment -Sodium Blood Sample Tests | Baseline to Day 360
  Changes from pre-dose value for Sodium (mEq/L)
Clinical laboratory assessment- Chloride Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Chloride (mmol/L)
Clinical laboratory assessment- Potassium Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Potassium (mEq/L)
Clinical laboratory assessment- Bicarbonate Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Bicarbonate (mEq/L)
Clinical laboratory assessment- Urea Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Urea mmol/L
Clinical laboratory assessment -Creatinine Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Creatinine (mg/dL)
Clinical laboratory assessment -Bilirubin (total) Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Bilirubin (mg/dL)
Clinical laboratory assessment -Bilirubin (direct) Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Bilirubin, direct only if total bilirubin is elevated (mg/dL)
Clinical laboratory assessment -Alkaline Phosphatase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Alkaline Phosphatase (U/L)
Clinical laboratory assessment -Aspartate aminotransferase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Aspartate aminotransferase (U/L)
Clinical laboratory assessment -Alanine aminotransferase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Alanine aminotransferase (U/L)
Clinical laboratory assessment -Lactate dehydrogenase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Lactate dehydrogenase (U/L)
Clinical laboratory assessment -Creatinine Kinase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Creatine kinase for (U/L)
Clinical laboratory assessment - Gamma glutamyl transferase Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Gamma glutamyl transferase (U/L)
Clinical laboratory assessment - Troponin Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Troponin (ng/mL)
Clinical laboratory assessment - Total Protein Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Total Protein (g/dL)
Clinical laboratory assessment - Albumin Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Albumin (g/dL)
Clinical laboratory assessment - Calcium Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Calcium (mg/dL)
Clinical laboratory assessment - Fasting Glucose Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Fasting Glucose (mg/dL)
Clinical laboratory assessment - Non Fasting Glucose Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Non Fasting Glucose (mg/dL)
Clinical laboratory assessment - Fasting Triglycerides Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Fasting Triglycerides (mg/dL)
Clinical laboratory assessment - Total Fasting Cholesterol Blood Sample Test | Baseline to Day 360
  Changes from pre-dose value for Total Fasting Cholesterol) (mg/dL)
Clinical laboratory assessment-Bilirubin Urine Sample Test | Baseline to Day 360
  Changes from pre-dose values for Bilirubin (mg/dL)
Clinical laboratory assessment-Urobilinogen Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Urobilinogen (mmol/L)
Clinical laboratory assessment- Ketones Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Ketones (mmol/L)
Clinical laboratory assessment- Glucose Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Glucose (mmol/L)
Clinical laboratory assessment- Protein Urine Sample Test | Baseline to Day 360
  Changes from pre-dose values for Protein (mg/dL)
Clinical laboratory assessment- Blood Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Blood (RBC/HPF)
Clinical laboratory assessment- Nitrites Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Nitrites (mg/dL)
Clinical laboratory assessment- pH Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for pH (pH value)
Clinical laboratory assessment- Specific Gravity Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Specific Gravity (USG)
Clinical laboratory assessment- Leukocytes Urine Sample Test | Baseline to Day 360
  Changes from pre-dose value for Leukocytes (leukocytes per microscopic field)
Clinical laboratory assessment- High Sensitivity C- Reactive Protein | Baseline to Day 360
  Changes from pre-dose value for High Sensitivity C- Reactive Protein (mg/L)

SECONDARY OUTCOMES:
Plasma PK Parameter of YCT-529 (Area under the curve to Infinity [AUCinf]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 extrapolated to infinity [AUCinf]
Plasma PK Parameter of YCT-529 (Area under the curve to the last measured concentration [AUC0-t]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 to the last measured concentration [AUC0-t]
Plasma PK Parameter of YCT-529 (Area under the curve to 24 hours [AUC0-24]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by area under the curve from time 0 to 24 hours [AUC0-24]
Plasma PK Parameter of YCT-529 (Time to maximum concentration [Tmax]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by time to maximum concentration [Tmax]
Plasma PK Parameter of YCT-529 (Terminal elimination half life [T1/2]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by terminal elimination half life [T1/2]
Plasma PK Parameter of YCT-529 (Lag time [Tlag]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by lag time [Tlag]
Plasma PK Parameter of YCT-529 (Volume of distribution [Vz/F]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by apparent volume of distribution [Vz/F]
Plasma PK Parameter of YCT-529 (oral clearance [CL/F]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by oral clearance [CL/F] of YCT-529
Plasma PK Parameter of YCT-529 (maximum concentration [Cmax]) | Pre-dose to 28 days and 90 days after dosing
  Plasma PK Parameter as measured by maximum concentration [Cmax]) of YCT-529
Pharmacodynamic parameter of YCT-529, including follicle-stimulating hormone | Pre-dose to 28 days and 90 days after dosing
  Changes from pre-dose values of follicle-stimulating hormone
Pharmacodynamic parameter of YCT-529, including luteinizing hormone | Pre-dose to 28 days and 90 days after dosing
  Changes from pre-dose values of luteinizing hormone
Pharmacodynamic parameter of YCT-529, including estradiol | Pre-dose to 28 days and 90 days after dosing
  Changes from pre-dose values of luteinizing hormone
Pharmacodynamic parameter of YCT-529, including testosterone | Pre-dose to 28 days and 90 days after dosing
  Changes from pre-dose values of testosterone
Changes in YCT-529 concentrations in semen | Pre-dose to 28 days and 90 days after dosing
  Changes in YCT-529 as measured by changes in serum concentrations in semen

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Katia, MBChB, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research (NZCR), Grafton, Auckland, New Zealand